CLINICAL TRIAL: NCT03464682
Title: Multi-center,Randomized,Double Blind, Double Dummy,Placebo Controlled, Efficacy and Safety Study of HS-25 in Combination With Atovastatin in Adults With Primary Hypercholesterolemia
Brief Title: Efficacy and Safety of HS-25 or in Combination With Atorvastatin in Chinese Adults With Primary Hypercholesterolemia
Acronym: HS-25-C-01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-25-C-01
Record Dates: First submitted 2018-02-07; First posted 2018-03-14 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-02

CONDITIONS: Primary Hypercholesterolemia
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- HS-25 10mg (Experimental): HS-25 10mg, Placebo of HS-25 1 tablet, Placebo of Aorvastatin 1 tablet, oral once daily, 12weeks
  Interventions: Drug: HS-25 10mg; Drug: Placebe of HS-25 and Atorvastatin
- HS-25 20mg (Experimental): HS-25 10mg 2 tablets, Placebo of Aorvastatin 1 tablet, oral once daily, 12weeks
  Interventions: Drug: HS-25 20mg; Drug: Placebe of HS-25 and Atorvastatin
- HS-25 10mg combination with Atorvastatin (Experimental): HS-25 10mg, Aorvastatin 10mg, Placebo of HS-25 1 tablet, oral once daily, 12 weeks
  Interventions: Drug: HS-25 10mg combination with Atorvastatin; Drug: Atorvastatin 10mg; Drug: Placebe of HS-25 and Atorvastatin
- HS-25 20mg combination with Atorvastatin (Experimental): HS-25 20mg, Aorvastatin 10mg, oral once daily, 12 weeks
  Interventions: Drug: HS-25 20mg combination with Atorvastatin; Drug: Atorvastatin 10mg
- Aorvastatin 10mg (Active Comparator): Aorvastatin 10mg, Placebo of HS-25 2 tablets, oral once daily, 12 weeks
  Interventions: Drug: Atorvastatin 10mg; Drug: Placebe of HS-25 and Atorvastatin
- Placebo of HS-25 and Aorvastatin (Placebo Comparator): Placebo of HS-25 2 tablets, Placebo of Aorvastatin 1 tablet, oral once daily, 12 weeks
  Interventions: Drug: Placebe of HS-25 and Atorvastatin

INTERVENTIONS:
Drug: HS-25 10mg — HS-25 10mg 1tablet add placebo of HS-25 1 tablet, placebo of Atorvastatin 1 tablet
  Arms: HS-25 10mg
Drug: HS-25 10mg combination with Atorvastatin — HS-25 10mg 1 tablet , Atorvastatin 10mg 1 tablet, Placebo of HS-25 1 tablet
  Arms: HS-25 10mg combination with Atorvastatin
Drug: HS-25 20mg combination with Atorvastatin — HS-25 10mg 2 tablets, Atorvastatin 10mg 1 tablet
  Arms: HS-25 20mg combination with Atorvastatin
Drug: Atorvastatin 10mg — Atorvastatin 10mg 1 tablet, placebo of HS-25 2 tablets
  Arms: Aorvastatin 10mg; HS-25 10mg combination with Atorvastatin; HS-25 20mg combination with Atorvastatin
Drug: HS-25 20mg — HS-25 10mg 2 tablets, placebo of Atorvastatin 1 tablet
  Arms: HS-25 20mg
Drug: Placebe of HS-25 and Atorvastatin — Placebe of HS-25 2 tablets, Placebo of Atorvastatin 1 tablets
  Arms: Aorvastatin 10mg; HS-25 10mg; HS-25 10mg combination with Atorvastatin; HS-25 20mg; Placebo of HS-25 and Aorvastatin

SUMMARY:
To determine the efficacy of the HS-25 (10mg or 20mg) or in combination with Atorvastatin (10mg)in reducing low density lipoprotein-cholesterol (LDL-C) levels after a 12-week period of treatment in adults with primary hypercholesterolemia; To determine the safety of HS-25 (10mg or 20mg) or in combination with Atorvastatin (10mg)in subjects with LDL-C after a 40-week period of treament.

DETAILED DESCRIPTION:
This is a 12-week, randomized, double-blind, double dummy, placebo-controlled study designed to assess the effects of the cholesterol absorption inhibitor HS-25 (10mg or 20mg) or in combination with Atorvastatin (10mg) on LDL-C levels in adults who have untreated LDL-C levels ranging from 3.36-4.88mmol/L(130-189 mg/dL)and fasting triglyceride levels < 350 mg/dL. Eligibility is restricted to 18-70 years old men or women who are using a highly effective birth control method or are not of childbearing potential;subjects with not treated by statins in six months before signature of the informed consent.Subjects with diabetes, a history of myocardial infarction or other clinical evidence of atherosclerotic vascular disease or treated are not eligible for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 18 to 70 years of age, male or female using a highly effective birth control method or not of child-bearing potential, at Visit 1 (screening visit);
* LDL-C 3.36mmol/L (130 mg/dL) to 4.88 mmol/L (189 mg/dL) (inclusive) on a cholesterol lowering diet but no lipid modifying drug treatment (statins) for at least 6 weeks before signed written informed consent;
* A qualifying LDL-C value must be obtained at the beginning and end of the placebo run-in (Visit 2 and Visit 3) and the Visit 3 value must be within 12% of the value at Visit 2, higher or lower; the average of both qualifying values must be in the range of 3.36mmol/L (130 mg/dL) to 4.88 mmol/L (189 mg/dL) (inclusive) for inclusion in the study.

Exclusion Criteria:

* Liver transaminases > 1.5 x upper limit of normal.
* Homozygous Familial Hypercholesterolemia.
* Subject who was diagnosed as diabetes with aged greater than 40 years old.
* Subject who was diagnosed as diabetes with one of the following of cardiovascular risk factorss: Hypertention Bp ≥ 140/90mmHg,or smoking, or low HDL-C (1.04mmol/L), or BMI≥28kg/m2.
* Women who are pregnant or breast feeding.
* Atherosclerotic cardiovascular disease including Arteriosclerotic heart disease, Acute coronary syndrome，Coronary artery bypass graft,Coronary angioplastyPeripheral arteriosclerosis,Cerebrovascular accident - history of Severe Endiocrine disease (for example Thyroid function abnormal) - History of a positive test for human immunodeficiency virus, hepatitis B or hepatitis C.
* History of advanced cancer - Arrhythmias need to be treated by medications
* Had severe injured or surgery in 6 months before study start.
* Hypersensitive to HS-25 or place.
* History of intolerance to ezetimibe.
* Participation other studies in three months.
* Treatment with a fibric acid derivative (eg, fenofibrate, gemfibrozil), probucol, warfarin, systemic corticosteroid, cyclosporine or other immunosuppressant agent within the prior 12 weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2015-02-28 (Actual); Primary Completion 2018-12-28 (Estimated); Study Completion 2019-05-28 (Estimated)

PRIMARY OUTCOMES:
Percent change of LDL-C | 12 weeks
  Percent change in LDL-C from baseline to week 12 for each group

SECONDARY OUTCOMES:
Percent change of LDL-C | 52 weeks ( including 2, 4, 8, 18, 24, 38, 52 weeks)
  Percent change in LDL-C from baseline to week 2, 4, 8, 18, 24, 38, 52 for each group
Percent change of Non-HDL-C | 52 weeks ( including 2, 4, 8, 12, 18, 24, 38, 52 weeks)
  Percent change in Non-HDL-C from baseline to week 2, 4, 8, 12, 18, 24, 38, 52 for each group
Percent change of HDL-C | 52 weeks ( including 2, 4, 8, 12, 18, 24, 38, 52 weeks)
  Percent change in HDL-C from baseline to week 2, 4, 8, 12, 18, 24, 38, 52 for each group
Percent change of TC, TG, Apo B, Apo Al | 52 weeks ( including 2, 4, 8, 12, 18, 24, 38, 52 weeks)
  Percent change in TC, TG, Apo B, Apo Al from baseline to week 2, 4, 8, 12, 18, 24, 38, 52 for each group

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University